CLINICAL TRIAL: NCT03299764
Title: Evaluation of Non-invasive Pursed-lip Breathing Ventilation (PLBV) in Advanced COPD
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Devices not available at the moment.
Sponsor: Research Center Borstel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZL PBLV Trial
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Non-invasive ventilation with pursed lip breathing ventilation device
  Interventions: Device: Pursed lip breathing ventilation
- Control (Active Comparator): Non-invasive ventilation with standard non-invasive ventilation device
  Interventions: Device: Standard non-invasive ventilation

INTERVENTIONS:
Device: Pursed lip breathing ventilation — A non-invasive ventilation device mimicking the pursed lip breathing in COPD patients will be used.
  Arms: Intervention
Device: Standard non-invasive ventilation — Standard non-invasive ventilation
  Arms: Control

SUMMARY:
Comparison of a conventional non-invasive ventilation to a non-invasive pursed-lip breathing ventilation (PLBV) ventilation in advanced COPD

DETAILED DESCRIPTION:
Intervention:

Non-invasive ventilation with dynamic positive pressure during expiration (pursed-lip breathing ventilation, PLBV) Control Conventional bi-level non-invasive ventilation (NIV) with static positive pressures Duration of intervention per patient 3 months as randomized (1:1) followed by 9 months as chosen by patient

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Age >40 years
3. COPD diagnosis known for at least 12 months
4. NIV therapy for at least 3 months

4. Regular use of NIV with extrapolated usage time of at least 700 hours / year 5. Current inspiratory NIV pressure ≥20 mbar 6. Patient understands the requirements of the study 7. Patient is able to follow the study protocol

Exclusion Criteria:

1. Current COPD exacerbation (is allowed 4 weeks after end of treatment)
2. Radiologically proven pneumonia within the past month
3. Other leading pulmonary illness
4. Tracheostomy
5. Pneumothorax
6. Pregnancy or lactation
7. BMI >35 kg/m²
8. Steroid therapy with >15 mg prednisolon daily for >1 month
9. Condition causing hypercapnia other than COPD
10. 6MWT distance of >300 meters within the last 7 days
11. Previous therapy with the Vigaro NIV device
12. Weight loss of more than 5 kg / 12 months
13. Further criteria to exclude confounding factors

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Walking distance in 6-minutes walking test | 3 months

SECONDARY OUTCOMES:
Mortality | 12 months
Number of hospital admissions | 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- Germany (5):
  - Thoraxklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Waldburg-Zeil Kliniken - Fachkliniken Wangen, Wangen, Baden-Wurttemberg
  - Research Center Borstel, Borstel, Schleswig-Holstein
  - LungenClinic Großhansdorf, Großhansdorf, Schleswig-Holstein
  - Lungenklinik Hemer, Hemer